CLINICAL TRIAL: NCT01473784
Title: A Pilot Study Assessing Transoral Robotic Surgery (TORS) for Oral and Laryngopharyngeal Benign and Malignant Lesions Using the Da Vinci Robotic Surgical System
Brief Title: Transoral Robotic Surgery in Treating Patients With Benign or Malignant Tumors of the Head and Neck
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Enver Ozer, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-07061; NCI-2011-03122 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2011-11-07; First posted 2011-11-17 (Estimated); Last update posted 2026-02-10 (Actual); Status verified 2026-01

CONDITIONS: Recurrent Adenoid Cystic Carcinoma of the Oral Cavity; Recurrent Mucoepidermoid Carcinoma of the Oral Cavity; Recurrent Squamous Cell Carcinoma of the Hypopharynx; Recurrent Squamous Cell Carcinoma of the Larynx; Recurrent Squamous Cell Carcinoma of the Lip and Oral Cavity; Recurrent Verrucous Carcinoma of the Larynx; Recurrent Verrucous Carcinoma of the Oral Cavity; Stage 0 Hypopharyngeal Cancer; Stage 0 Laryngeal Cancer; Stage 0 Lip and Oral Cavity Cancer; Stage I Adenoid Cystic Carcinoma of the Oral Cavity; Stage I Mucoepidermoid Carcinoma of the Oral Cavity; Stage I Squamous Cell Carcinoma of the Hypopharynx; Stage I Squamous Cell Carcinoma of the Larynx; Stage I Squamous Cell Carcinoma of the Lip and Oral Cavity; Stage I Verrucous Carcinoma of the Larynx; Stage I Verrucous Carcinoma of the Oral Cavity; Stage II Adenoid Cystic Carcinoma of the Oral Cavity; Stage II Mucoepidermoid Carcinoma of the Oral Cavity; Stage II Squamous Cell Carcinoma of the Hypopharynx; Stage II Squamous Cell Carcinoma of the Larynx; Stage II Squamous Cell Carcinoma of the Lip and Oral Cavity; Stage II Verrucous Carcinoma of the Larynx; Stage II Verrucous Carcinoma of the Oral Cavity; Stage III Adenoid Cystic Carcinoma of the Oral Cavity; Stage III Mucoepidermoid Carcinoma of the Oral Cavity; Stage III Squamous Cell Carcinoma of the Hypopharynx; Stage III Squamous Cell Carcinoma of the Larynx; Stage III Squamous Cell Carcinoma of the Lip and Oral Cavity; Stage III Verrucous Carcinoma of the Larynx; Stage III Verrucous Carcinoma of the Oral Cavity; Stage IV Squamous Cell Carcinoma of the Hypopharynx; Stage IVA Adenoid Cystic Carcinoma of the Oral Cavity; Stage IVA Mucoepidermoid Carcinoma of the Oral Cavity; Stage IVA Squamous Cell Carcinoma of the Larynx; Stage IVA Squamous Cell Carcinoma of the Lip and Oral Cavity; Stage IVA Verrucous Carcinoma of the Larynx; Stage IVA Verrucous Carcinoma of the Oral Cavity; Stage IVB Adenoid Cystic Carcinoma of the Oral Cavity; Stage IVB Mucoepidermoid Carcinoma of the Oral Cavity; Stage IVB Squamous Cell Carcinoma of the Larynx; Stage IVB Squamous Cell Carcinoma of the Lip and Oral Cavity; Stage IVB Verrucous Carcinoma of the Larynx; Stage IVB Verrucous Carcinoma of the Oral Cavity; Stage IVC Adenoid Cystic Carcinoma of the Oral Cavity; Stage IVC Mucoepidermoid Carcinoma of the Oral Cavity; Stage IVC Squamous Cell Carcinoma of the Larynx; Stage IVC Squamous Cell Carcinoma of the Lip and Oral Cavity; Stage IVC Verrucous Carcinoma of the Larynx; Stage IVC Verrucous Carcinoma of the Oral Cavity; Tongue Cancer
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Hypopharyngeal Neoplasms; Laryngeal Neoplasms; Mouth Neoplasms; Tongue Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Transoral robotic surgery (TORS) (Experimental): Patients will undergo TORS for oral and laryngopharyngeal benign and malignant lesions using the Da Vinci Robotic Surgical System. After surgery regular clinical assessments will be scheduled to see how the patient is doing. Patients will be asked to answer a quality of life assessment as part of the study. If patients are unable to come to the Ohio State University Medical Center for a physician appointment they will be contacted via phone or mailed a questionnaire to complete.
  Interventions: Procedure: transoral robotic surgery; Procedure: quality of life assessment

INTERVENTIONS:
Procedure: transoral robotic surgery — Undergo TORS using the Da Vinci Robotic Surgical System
  Other Names: TORS; DA VINCI® ROBOTIC SURGICAL SYSTEM
Procedure: quality of life assessment — After surgery regular clinical assessments will be scheduled to see how the patient is doing. Patients will be asked to answer a quality of life assessment as part of the study. If patients are unable to come to the Ohio State University Medical Center for a physician appointment they will be contacted via phone or mailed a questionnaire to complete.
  Other Names: questionnaire

SUMMARY:
This pilot clinical trial studies transoral robotic surgery (TORS) in treating patients with benign or malignant tumors of the head and neck. TORS is a less invasive type of surgery for head and neck cancer and may have fewer side effects and improve recovery

DETAILED DESCRIPTION:
To conduct a pilot single-arm study to assess transoral robotic surgery (TORS) for oral and laryngopharyngeal benign and malignant lesions using the Da Vinci Robotic Surgical System.

ELIGIBILITY:
Inclusion Criteria:

* Patient must present with indications for diagnostic or therapeutic approaches for benign and/or malignant diseases of the oral cavity or laryngopharynx (including the neoplastic lesions of the tongue, tongue base, retromolar trigone, tonsils, palate, posterior and lateral pharynx, glottic, supraglottic and subglottic larynx)
* Patients must have adequate transoral exposure of the oral cavity and laryngopharynx for TORS instrumentation
* Written informed consent and/or Consent waiver by institutional review board (IRB)

Exclusion Criteria:

* Unexplained fever and/or untreated, active infection
* Patient pregnancy
* Previous head and neck surgery that would preclude transoral/robotic procedures. This is at the investigator's discretion. This is not an exclusion criterion for the non-surgical arm.
* The presence of medical conditions contraindicating general anesthesia or transoral surgical approaches
* Inability to grant informed consent
* INTRAOPERATIVE EXCLUSION CRITERIA:
* Inability to adequately visualize anatomy to perform the diagnostic or therapeutic surgical approach transorally

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2007-12-03 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Determine the feasibility of the TORS in patients with oral and laryngopharyngeal benign and malignant lesions. | up to eight years

SECONDARY OUTCOMES:
Assess the impact of TORS on the intra-operative surgical outcomes such as operative time, blood loss and complications. | up to eight years
  If the planned procedure is a combined procedure, (robotic + non robotic) above mentioned measures are going to be presented separately for successful fully robotic surgeries and for unsuccessful mixed surgeries.
  2. To identify the learning curve for TORS by measuring the efficiency and accuracy of the surgeons who perform the procedures.
Assess the quality of life of the patients with TORS. | up to eight years

CONTACTS AND LOCATIONS:
Overall Officials: Enver Ozer, MD, Principal Investigator — Ohio State University
Locations (1):
- Ohio State University Medical Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Jamesline — http://cancer.osu.edu